CLINICAL TRIAL: NCT03812107
Title: Response to Relapse in Office-Based Opioid Treatment Trial
Acronym: RR-OBOT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to COVID-19 as it interfered with the study intervention.
Sponsor: Boston Medical Center (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-38177; 1H79TI081600-01 (Other Grant/Funding Number: Substance Abuse and Mental Health Services Administration)
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Opioid-use Disorder
Keywords: Opioid-use Disorder (OUD); Medication for OUD (MOUD); Co-occurring opioid use disorder and mental disorders; Office-based Addiction Treatment
MeSH Terms: conditions — Opioid-Related Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Treatment Approach (Experimental): Participants in this arm who relapse will be able to move more freely between follow up steps and are hypothesized to require fewer provider visits than those in the intensive treatment arm.
  Interventions: Other: Moderate Treatment Approach
- Intensive Treatment Approach (Active Comparator): Participants in this arm who relapse will follow the current guidelines follow up steps of weekly, then every two weeks and finally monthly provider visits.
  Interventions: Other: Intensive Treatment Approach

INTERVENTIONS:
Other: Moderate Treatment Approach — The frequency of visits will be organized similarly as the intensive treatment arm (weekly, every 2 weeks, and every 4 weeks) but participants in this arm will be able to move more freely between these steps and are hypothesized to require fewer provider visits than the intensive treatment arm.
  Arms: Moderate Treatment Approach
Other: Intensive Treatment Approach — After stabilization on a MOUD, participants who relapse will be asked to return weekly until 2 consecutive urine drug tests are negative for opioids or other illicit drugs. Participants will then be asked to return every other week until 2 consecutive urine drug tests are negative for opioids or other illicit drugs, before being asked to return every 4 weeks. If the participant tests positive for illicit drugs while returning every other week, they will return to the beginning of the treatment plan (2 consecutive negative tests before going to every other week).
  Arms: Intensive Treatment Approach

SUMMARY:
In a sample of individuals with co-occurring OUD and mental disorders, the investigators plan to test two medications for opioid use disorder (MOUD) treatment protocols that involve differing approaches to the use of opioids and other drugs during and after stabilization on MOUD - intensive vs. moderate treatment.The study is being conducted alongside the opening of a new clinical service funded by the Substance Abuse and Mental Health Services Administration (SAMHSA) known as the Addiction and Behavioral Health Outpatient Recovery (ABOVE) program. The ABOVE Program is designed to treat patients with co-occurring opioid use disorder (OUD) and mental disorders with MOUD. Participants are individuals seeking treatment for co-occurring opioid use disorder (OUD) and mental disorders and are willing to receive MOUD treatment. Potential participants will be screened in the context of clinical care for opioid use disorder and mental disorders. If they are eligible for treatment in the ABOVE program, they will be asked to complete a baseline assessment, again for the purposes of clinical care. After completing the baseline clinical assessment, they will be asked to participate in this clinical trial, consented, then randomized. Treatment is delivered in the context of clinical care which involves delivery of MOUD and can involve psychiatric medications, and group and individual psychotherapy. Difference in treatment between the two randomization arms will only occur if a relapse to drug use occurs and will only involve two protocol-directed treatment responses to relapse.

DETAILED DESCRIPTION:
This study is a single-center, two-arm, 6-month (24-week), parallel group, open-label, randomized controlled trial to examine the effectiveness of two approaches to managing relapse to illicit drug use in treatment with medications for opioid use disorder (MOUD). It will compare two treatment protocols for treatment of opioid use disorder with medications. The two protocols involve differing approaches to relapse to use of illicit drugs in a sample of individuals with co-occurring OUD and mental disorders.

Intensive Treatment Approach: After stabilization on a medication for OUD (MOUD), if a participant tests positive for opioids or other illicit drugs, they will be asked to return weekly until 2 consecutive urine drug tests are negative for opioids or other illicit drugs. Participants will then be asked to return every other week until 2 consecutive urine drug tests are negative for opioids or other illicit drugs, before being asked to return every 4 weeks. If the participant tests positive for illicit drugs while returning every other week, they will return to the beginning of the treatment plan (2 consecutive negative tests before going to every other week).

Moderate treatment approach: The frequency of visits will be organized similarly as the intensive treatment arm (weekly, every 2 weeks, and every 4 weeks) but participants in this arm will be able to move more freely between these steps and are hypothesized to require fewer provider visits than the intensive treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Opioid use disorder [based on Diagnostic Statistical Manual 5 (DSM5) criteria assessed by clinician interview]
* Mental disorder (based on DSM5 criteria assessed by clinician interview)
* Willingness to receive treatment with office-based medication for opioid use disorder
* Willingness to name at least 1 contact for follow up purposes
* Enrollment in the ABOVE program

Exclusion Criteria:

* Pregnancy (urine testing if childbearing potential) or breast feeding
* Suicidal or homicidal ideation that requires immediate attention
* Cognitive dysfunction that precludes informed consent or research staff assessment that participant cannot understand interview questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Retention in MOUD treatment | 24 weeks
  This is a continuous measure of days a participant is prescribed medications for opioid use disorder for 24 weeks. For example, if the first prescription is for 7 days, then this measure has a minimum value of 7 days and a maximum value of approximately 168 days (24 weeks). If a participant is without MOUD prescribed by the ABOVE clinical program for 7 days or greater, then the participant will be considered discontinued from treatment for study purposes.

SECONDARY OUTCOMES:
Number of medications for opioid use disorder provider visits | 24 weeks
  The number of provider visits attended will be recorded for each participant. Types of provider visits include visits with a nurse, psychiatrist, nurse practitioner, or mental health clinician for either individual or group psychotherapy.
Change in number of days of past 30-day illicit opioid use by self-report from baseline to 24 weeks | baseline, 24 weeks
  Participants will be asked the number of days of illicit opioid use (includes use of non-prescribed opioid analgesics) in the past 30 days at baseline and 24 week follow-up. This outcome will be the difference in the number of days of illicit opioid use between baseline and 24 weeks.
Change in number of days of past 30-day any illicit drug use or heavy drinking days by self-report from baseline to 24 weeks | baseline, 24 weeks
  Participants will be asked the number of days of any illicit drug use or heavy drinking days (5 or more alcoholic drinks in one sitting for males or 4 or more alcohol drinks in one sitting for females) in the past 30 days at baseline and 6 month follow-up. This outcome will be the difference in the number of days of any illicit drug use or heavy drinking days between baseline and 6 months.
Proportion of urine drug tests negative for opioids from baseline to 24 weeks | 24 weeks
  Participants will be asked to provide urine drug tests that test for illicit drugs including illicit opioids at least once every 4 weeks from baseline to 24 weeks. Because urine drug tests will only be obtained on clinical visit days and the two arms may have a different number of urine drug tests obtained per participant, only monthly or near-monthly drug tests in each arm (week 4, week 8, week 12, etc.) will be included in the study.
Proportion of urine drug tests negative for any illicit drug from baseline to 24 weeks | 24 weeks
  Participants will be asked to provide urine drug tests that test for illicit drugs including amphetamines, barbiturates, cocaine, benzodiazepines, opioids (including opiates, fentanyl, oxycodone, methadone), at least once every 4 weeks from baseline to 24 weeks. Because urine drug tests will only be obtained on clinical visit days and the two arms may have a different number of urine drug tests obtained per participant, only monthly or near-monthly drug tests in each arm (week 4, week 8, week 12, etc.) will be included in the study.
Participant satisfaction using the TPQ | 24 weeks
  The Treatment Perceptions Questionnaire (TPQ) is a 10-item questionnaire with Likert scale responses from 0 to 4 it also allows open-responses / feedback. Potential range of scores is from 0 to 40 and higher scores indicate greater satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Christina Borba, PhD MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT03812107/ICF_000.pdf